CLINICAL TRIAL: NCT02268175
Title: A Phase II Randomized Study of Enzalutamide+Leuprolide Versus Enzalutamide+Leuprolide+Abiraterone Acetate+Prednisone as Neoadjuvant Therapy for HIgh-Risk Prostate Cancer Undergoing Prostatectomy
Brief Title: Enzalutamide/Leuprolide +/- Abiraterone/Pred in Prostate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Principal Investigator, Mary-Ellen Taplin, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-283
Record Dates: First submitted 2014-10-14; First posted 2014-10-20 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-03

CONDITIONS: Prostate Adenocarcinoma; Prostate Cancer; High Risk Prostate Cancer
Keywords: prostate adenocarcinoma; advanced prostate cancer; high risk prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; Abiraterone Acetate; Prednisone; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM 1 (Experimental): Participants will be randomized in a 2:1 ratio to neoadjuvant treatment (ARM 1) or (ARM 2).
  Participants will receive the assigned study treatment per cycle
  * Enzalutamide- Once daily at prespecified dose, orally
  * Abiraterone Acetate- Once daily at prespecified dose, orally
  * Prednisone-Once daily at prespecified dose, orally
  * Leuprolide Acetate-Intermuscular injection at prespecified dose and duration
  Interventions: Drug: Enzalutamide; Drug: Abiraterone Acetate; Drug: Prednisone; Drug: Leuprolide Acetate
- ARM 2 (Experimental): Participants will be randomized in a 2:1 ratio to neoadjuvant treatment (ARM 1) or (ARM 2).
  Participants will receive the assigned study treatment per cycle.
  * Enzalutamide- once daily at prespecified dose, orally
  * Leuprolide Acetate- Intermuscular injection at prespecified dose and duration
  Interventions: Drug: Enzalutamide; Drug: Leuprolide Acetate

INTERVENTIONS:
Drug: Enzalutamide — 160 mg (four 40 mg capsules), oral, once daily, 28 days (4 weeks) 6 cycles maximum. Can be taken with or without food.
  Other Names: XTANDI
Drug: Abiraterone Acetate — 1000 mg (four 250 mg tablets), oral, once daily, 28 days (4 weeks) 6 cycles maximum. No food should be consumed for at least two hours before the dose and for at least one hour after the dose.
  Other Names: Zytiga
  Arms: ARM 1
Drug: Prednisone — 5 mg, oral, once daily, 28 days (4 weeks) 6 cycles maximum.Take with food, preferred to be taken in the morning .
  Arms: ARM 1
Drug: Leuprolide Acetate — Either 7.5 mg monthly or 22.5 mg every three months, Intramuscular, monthly or every three months.
  Other Names: - Lupron Depot-3 Month; - Lupron Depot-4 Month; - Lupron Depot; - Lupron; - Viadur

SUMMARY:
This study is comparing the effectiveness of enzalutamide with or without abiraterone acetate for men with high-risk, localized prostate cancer.

DETAILED DESCRIPTION:
In this research study, the investigators are comparing the effectiveness of enzalutamide with or without abiraterone acetate for men with high-risk, localized prostate cancer.

Abiraterone acetate with prednisone and enzalutamide are currently FDA-approved for use in the treatment of patients with metastatic castration-resistant prostate cancer, however they are investigational for the treatment of localized prostate cancer. Abiraterone acetate works by decreasing the production of male sex hormones, which cause prostate cancer growth. Enzalutamide works by blocking the effects of male sex hormones, which cause prostate cancer growth.

The FDA (the U.S. Food and Drug Administration) has not approved the combination of enzalutamide and abiraterone acetate as neoadjuvant therapy for high risk prostate cancer undergoing prostatectomy but each drug has been approved for the treatment of more advanced prostate cancer.

Participants will be randomized to one of two study arms. Randomization means that the participant is put into a group by chance. It is like flipping a coin. Neither participant nor the research doctor will choose what group participants are randomized to.

The names of the study medications involved in this study are:

* Enzalutamide
* Abiraterone Acetate
* Prednisone
* Leuprolide Acetate

ELIGIBILITY:
Inclusion Criteria:

* Male greater than or equal 18 years of age.
* Histologically confirmed adenocarcinoma of the prostate without histological variants (including overt neuroendocrine differentiation, small cell neuroendocrine carcinoma features, sarcomatoid features, pure ductal adenocarcinoma, squamous or transitional cell carcinoma).
* Must have tissue available from the pre-treatment diagnostic biopsy (tissue blocks if possible; if not possible, 10 unstained slides from each positive core sample for a total of 30 slides).
* Must have three core biopsies involved with cancer (a minimum of 6 core biopsies must be obtained). Prostate biopsy must be within three months from screening.
* Participants must have the following features:

  * Intermediate-risk disease defined as Gleason 4+3=7 disease OR
  * High-risk disease defined as Gleason 8-10 OR PSA > 20 ng/dL OR T3 disease (by prostate MRI)
* No evidence of metastatic or nodal disease as determined by radionuclide bone scans CT/MRI.
* Participants must be candidates for RP and considered surgically resectable by urologic evaluation.
* ECOG performance status 0 to 1 (Appendix A).
* Participants must have normal organ and marrow function as defined below:

  * WBC ≥ 3,000/mcL
  * ANC ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Serum potassium ≥ 3.5 mmol/L
  * AST, ALT, and total bilirubin ≤ 1.5 x Institutional ULN
  * Calculated creatinine clearance ≥ 60 mL/min
  * PTT ≤ 60, INR ≤ 1.5 x Institutional ULN unless on warfarin therapy (investigator would need to determine if safe for participant to stop warfarin prior to biopsy and warfarin therapy)
  * Controlled blood pressure defined as a systolic blood pressure ≤ 140 mmHg and diastolic blood pressure ≤ 90 mmHg on no more than three anti-hypertensive agents. Drug formulations containing two or more anti-hypertensive agents will be counted based on the number of active agents in each formulation.

Exclusion Criteria:

* Prior hormone therapy for prostate cancer including orchiectomy, antiandrogens (including first-generation antiandrogens, enzalutamide, ARN-509 and others), CYP17 inhibitors (including abiraterone, TAK-700, galeterone, ketoconazole, and others), estrogens, LHRH agonist/antagonists. Prior therapy with 5α-reductace inhibitors is allowed. LHRH therapy allowed if begun within 4 weeks of day 1.
* Prior chemotherapy, radiation therapy, or immunotherapy for prostate cancer.
* Prior systemic treatment with an azole drug within four weeks of screening visit.
* Hypogonadism or severe androgen deficiency as defined by screening serum testosterone < 200 ng/dL.
* Clinically significant cardiovascular disease including:
* Acute coronary syndrome within 6 months of screening visit;

  * Hypotension defined as a systolic blood pressure < 86 mmHg;
  * Bradycardia defined as a heart rate of < 50 beats per minute, unless pharmaceutically induced and thus reversible (i.e. beta blockers);
  * Uncontrolled angina (requiring escalating doses of nitrates) within 3 months of screening visit;
  * Congestive heart failure NYHA Class III or IV or subjects with a history of congestive heart failure NYHA Class III or IV, unless screening ECHO results in left ventricular ejection fraction that ≥ 45%;
  * History of clinically significant ventricular arrhythmias (e.g. ventricular tachycardia, ventricular fibrillation, torsades de pointes);
  * Prolonged corrected QT interval by the Fridericia correction formula (QTcF) on screening EKG > 470 msec;
  * History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place;
* History of seizure or any condition or concurrent medication that may predispose to seizure.
* Thromboembolism within 6 months of screening visit.
* Severe hepatic impairment (Child-Pugh Class C).
* Active or symptomatic viral hepatitis or chronic liver disease.
* History of pituitary or adrenal dysfunction.
* GI disorders which may interfere with the absorption of the study drug.
* Pre-existing condition that warrants long-term corticosteroid use.
* Concomitant use of medications that may alter pharmacokinetics of abiraterone or enzalutamide.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances: 1) individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy, or 2) individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: non-muscle invasive bladder cancer, basal cell or squamous cell carcinoma of the skin.
* Major surgery or radiation therapy within 30 days of screening.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-10; Primary Completion 2018-01 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Ellen Taplin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Johns Hopkins University, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] McKay RR, Ye H, Xie W, Lis R, Calagua C, Zhang Z, Trinh QD, Chang SL, Harshman LC, Ross AE, Pienta KJ, Lin DW, Ellis WJ, Montgomery B, Chang P, Wagner AA, Bubley GJ, Kibel AS, Taplin ME. Evaluation of Intense Androgen Deprivation Before Prostatectomy: A Randomized Phase II Trial of Enzalutamide and Leuprolide With or Without Abiraterone. J Clin Oncol. 2019 Apr 10;37(11):923-931. doi: 10.1200/JCO.18.01777. Epub 2019 Feb 27. PMID 30811282

RESULTS

PARTICIPANT FLOW:
Groups:
- Enzalutamide + Abiraterone + Prednisone + Leuprolide: Enzalutamide: 160 mg (four 40 mg capsules), oral, once daily, 28 days (4 weeks) 6 cycles maximum.
  Abiraterone Acetate: 1000 mg (four 250 mg tablets), oral, once daily, 28 days (4 weeks) 6 cycles maximum.
  Prednisone: 5 mg, oral, once daily, 28 days (4 weeks) 6 cycles maximum.
  Leuprolide Acetate: Either 7.5 mg monthly or 22.5 mg every three months, Intramuscular, monthly or every three months.
- Enzalutamide + Leuprolide: Enzalutamide: 160 mg (four 40 mg capsules), oral, once daily, 28 days (4 weeks) 6 cycles maximum.
  Leuprolide Acetate: Either 7.5 mg monthly or 22.5 mg every three months, Intramuscular, monthly or every three months.
Period: Overall Study
Arm/Group | Enzalutamide + Abiraterone + Prednisone + Leuprolide | Enzalutamide + Leuprolide
Started | 50 | 25
Completed | 50 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ARM 1: Enzalutamide: 160 mg (four 40 mg capsules), oral, once daily, 28 days (4 weeks) 6 cycles maximum.
  Abiraterone Acetate: 1000 mg (four 250 mg tablets), oral, once daily, 28 days (4 weeks) 6 cycles maximum.
  Prednisone: 5 mg, oral, once daily, 28 days (4 weeks) 6 cycles maximum.
  Leuprolide Acetate: Either 7.5 mg monthly or 22.5 mg every three months, Intramuscular, monthly or every three months.
- ARM 2: Enzalutamide: 160 mg (four 40 mg capsules), oral, once daily, 28 days (4 weeks) 6 cycles maximum.
  Leuprolide Acetate: Either 7.5 mg monthly or 22.5 mg every three months, Intramuscular, monthly or every three months.
- Total: Total of all reporting groups
Arm/Group | ARM 1 | ARM 2 | Total
Number analyzed (Participants) | 50 | 25 | 75
Age, Continuous [Median (Full Range); unit: years] | 62 [44 to 75] | 63 [52 to 73] | 62 [44 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 50 | 25 | 75
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 45 | 20 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
National Comprehensive Cancer Network (NCCN) Risk Group [Count of Participants; unit: Participants] — NCCN defined high risk: Gleason score>/=8, or prostate specific antigen (PSA)>20 ng/mL, or clinical stage T3 (tumor extends through prostate capsule or involves structures other than seminal vesicles) or higher and intermediate risk: Gleason score 4+3=7 disease
  Participants
    High Risk | 44 | 21 | 65
    Intermediate Risk | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pathologic Complete Response (pCR) or Minimal Residual Disease (MRD)
Description: pCR is defined as the absence of morphologically identifiable carcinoma in the radical prostatectomy (RP) specimen. MRD is defined as the largest cross-sectional dimension of residual tumor measuring </= 0.5 cm. If the tumor is multifocal, the size of the largest focus will be used to determine the size of the residual tumor.
Time Frame: after RP approximately 24 weeks from study entry
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ARM 1 | ARM 2
Number analyzed (Participants) | 50 | 25
percentage of participants | 30 [18 to 45] | 16 [5 to 36]
Statistical Analysis 1: Comparison: ARM 1 vs ARM 2; The hypothesis was that treatment with ARM 1 will have a pCR/MRD rate of 35% compared with Arm 2 rate of 10%. Given 75 men randomized in 2:1 ratio to Arm 1 (N=50) or Arm 2 (N=25), there was 84% power to detect this difference, using Fisher's exact test with one-sided type I error of 0.1; Test type: Superiority; p = 0.151, Fisher Exact — 1-sided

2. Secondary Outcome: Participants With Pathologic Complete Response (pCR)
Description: pCR is defined as the absence of morphologically identifiable carcinoma in the radical prostatectomy (RP) specimen.
Time Frame: after RP approximately 24 weeks from study entry
Measure: Count of Participants; unit: Participants
Arm/Group | ARM 1 | ARM 2
Number analyzed (Participants) | 50 | 25
Participants | 5 | 2

3. Secondary Outcome: Residual Cancer Burden (RCB)
Description: RCB was analyzed using radical prostatectomy (RP) tissue. The largest area of tumor was measured by ruler and the longest tumor dimension in this area was used as the dimension for calculation.
Time Frame: after RP approximately 24 weeks from study entry
Measure: Median (Full Range); unit: cm
Arm/Group | ARM 1 | ARM 2
Number analyzed (Participants) | 50 | 25
cm | 0.03 [0.0 to 4.0] | 0.05 [0.0 to 5.0]

4. Secondary Outcome: Positive Surgical Margin Status
Description: Participants were classified by presence or absence of positive surgical margins defined as margins, which are the edges of the removed tumor, that show some cancer cells.
Time Frame: after RP approximately 24 weeks from study entry
Measure: Count of Participants; unit: Participants
Arm/Group | ARM 1 | ARM 2
Number analyzed (Participants) | 50 | 25
Participants
  Absence | 41 | 22
  Presence | 9 | 3

5. Secondary Outcome: Median Prostate Specific Antigen (PSA) Nadir
Description: PSA nadir is the lowest PSA level recorded during neoadjuvant therapy.
Time Frame: PSA was assessed at baseline and every cycle during neoadjuvant therapy (up to 24 weeks).
Measure: Median (Full Range); unit: ng/mL
Arm/Group | ARM 1 | ARM 2
Number analyzed (Participants) | 50 | 25
ng/mL | 0.03 [0.0 to 0.27] | 0.02 [0.0 to 0.14]

ADVERSE EVENTS:
Time Frame: Assessed over treatment duration of 24 weeks.
Arm/Group | ARM 1 | ARM 2
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/25
Serious Adverse Events (participants affected / at risk) | 3/50 | 1/25
Other Adverse Events (participants affected / at risk) | 50/50 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARM 1 (N=50) | ARM 2 (N=25)
Pain (General disorders) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0
Hematoma (Vascular disorders) | 1 | 0
Cardiac disorders - Other (Cardiac disorders) | 0 | 1
Hot flashes (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARM 1 (N=50) | ARM 2 (N=25)
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Alanine aminotransferase increased (Investigations) | 17 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 16 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Bladder infection (Infections and infestations) | 1 | 0
Blood bilirubin increased (Investigations) | 2 | 1
Blurred vision (Eye disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cholesterol high (Investigations) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0
Concentration impairment (Nervous system disorders) | 0 | 2
Confusion (Psychiatric disorders) | 2 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 3
Diarrhea (Gastrointestinal disorders) | 2 | 0
Dizziness (Nervous system disorders) | 3 | 1
Dry eye (Eye disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 1 | 2
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 0 | 1
Endocrine disorders - Other (Endocrine disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 3 | 2
Eye disorders - Other (Eye disorders) | 0 | 1
Fatigue (General disorders) | 32 | 16
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 0
General disorders and administration site conditions - Other (General disorders) | 2 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 3
Gynecomastia (Reproductive system and breast disorders) | 4 | 0
Gynecomastia (Reproductive system and breast disorders) | 0 | 3
Hallucinations (Psychiatric disorders) | 1 | 0
Headache (Nervous system disorders) | 6 | 0
Headache (Nervous system disorders) | 0 | 3
Hematuria (Renal and urinary disorders) | 2 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hot flashes (Vascular disorders) | 41 | 22
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 17 | 7
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 | 2
Hypokalemia (Metabolism and nutrition disorders) | 5 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Infusion related reaction (General disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 9 | 0
Insomnia (Psychiatric disorders) | 0 | 4
Investigations - Other (Investigations) | 2 | 0
Irritability (General disorders) | 2 | 1
Lethargy (Nervous system disorders) | 1 | 0
Libido decreased (Psychiatric disorders) | 5 | 4
Memory impairment (Nervous system disorders) | 5 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 5 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 4 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Nervous system disorders - Other (Nervous system disorders) | 3 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 6 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Papulopustular rash (Infections and infestations) | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 0
Presyncope (Nervous system disorders) | 0 | 1
Psychiatric disorders - Other (Psychiatric disorders) | 6 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 4 | 5
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 3 | 2
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Restlessness (Psychiatric disorders) | 0 | 2
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 4 | 1
Skin infection (Infections and infestations) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Testicular disorder (Reproductive system and breast disorders) | 1 | 1
Tooth development disorder (Gastrointestinal disorders) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 3 | 1
Urinary frequency (Renal and urinary disorders) | 6 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Urinary urgency (Renal and urinary disorders) | 2 | 1
Vascular disorders - Other (Vascular disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Weight loss (Investigations) | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
White blood cell decreased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT02268175/Prot_SAP_000.pdf